CLINICAL TRIAL: NCT06263166
Title: The Effect of Using a Stress Ball During Vaginal Examination on Anxiety and Pain Levels
Brief Title: The Effect of Using a Stress Ball During Vaginal Examination on Anxiety and Pain Levels: a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nedime Gul Dogan Ozdemir, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5535
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Anxiety State; Pain; Exanimation
MeSH Terms: conditions — Anxiety Disorders; Pain; Coma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): No intervention other than usual care
- Intervention group (Experimental): Received stress ball intervention and usual care
  Interventions: Behavioral: Stress ball intervention

INTERVENTIONS:
Behavioral: Stress ball intervention — Women should squeeze and loosen the stress ball given to them during the vaginal examination and continue this process until the examination is completed.
  Arms: Intervention group

SUMMARY:
Women who will undergo vaginal examinations randomly assigned to intervention (n = 44) and control (n = 44) groups at a public hospital in Turkey will participate in the study. Stress ball application before vaginal examination will be explained to women in the intervention group. These women will be asked to tighten and loosen the stress ball given to them during the vaginal examination and continue this process until the examination is completed. Data regarding pain and anxiety outcomes will be collected before and after the examination.

The main questions it aims to answer are:

* question 1: What is the effect of stress ball application on women's anxiety level during vaginal examination?
* question 2: What is the effect of stress ball application on women's pain level during vaginal examination?

DETAILED DESCRIPTION:
Although vaginal examinations take less time than all other medical interventions, they create anxiety and negative thoughts in women. However, the vaginal examination has an important place in women's health as it helps detect sexually transmitted diseases, oncological processes, and all other changes early. Women shy away from gynecological examinations or postpone the examination due to the meanings they attach to gynecological examination and their physical or psychological negative experiences. This situation causes changes in the woman's health not to be detected early and to the emergence of negative consequences. For this reason, vaginal examination should not be performed in a way that increases the woman's anxiety, and methods that will facilitate the examination process should be used . Women state that they feel defenseless and that they hand over complete control to the person examining their reproductive organs, which they prefer to share only with their sexual partners . In a study evaluating the degree of physical discomfort during gynecological examination on a scale from 0 to 10, women defined the pain they experienced as six or more points. Other studies report that women have a more positive experience when techniques such as relaxation exercises, listening to music, or aromatherapy are used before or during vaginal examination. In addition to these techniques, visual, auditory, or tactile stimuli can focus women in a calmer state. Tactile stimuli, in particular, have the most effortless and natural potential for reducing anxiety or pain. The stress ball, one of the tactile stimuli, is thought to be an easy-to-use, non-invasive, non-pharmacological, inexpensive, and easily accessible method that helps the person focus elsewhere by distracting attention. Healthcare professionals need to reduce people's anxiety and ensure their comfort by developing positive coping mechanisms. Especially during the vaginal examination process, which is considered private in society, the majority of women expect nurses to be understanding and gentle and to know the methods that will make the woman feel comfortable. Lavender oil, one of the non-pharmacological applications during vaginal examination, has been shown to reduce anxiety and pain, and studies are comparing its positive effect. However, there is a need to investigate this, as there are no studies investigating the effectiveness of non-pharmacological methods of vaginal examination, especially the stress ball. No studies have been found. Although there are studies in the literature investigating the effectiveness of the stress ball, one of the non-pharmacological methods, in the treatment of various disease groups and symptoms , vaginal examination. No study has been found examining the effectiveness of a stress ball during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Those between the ages of 18-65,
* Applying to the polyclinic for vaginal examination,
* It is planned to recruit women who can read and write Turkish.

Exclusion Criteria:

* Pregnant,
* Having a diagnosed psychiatric problem such as depression, anxiety disorder, panic attack, bipolar affective disorder or schizophrenia
* It is planned to exclude women with visual, hearing, speech, physical, or mental disabilities.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Anxiety change | Immediately after the intervention
  As assessed by the State-Trait Anxiety Inventory (STAI) STAI consists of two scales, a total of 40 self-reported items. The State Anxiety Scale only used in this study, consists of 20 straight and inverse scored terms, and is scored between 20 and 80 in a likert type scoring between 1 and 4. High scores indicate high anxiety levels.
Pain level | Immediately after the intervention
  Visual Analog Scale (VAS) will be used to determine the severity of pain experienced by women in the intervention and control groups during vaginal examination. VAS converts values that cannot be measured numerically into numerical values. This scale is widely used for pain assessment. The pain level varies between 0 and 10, and an increase in the marked numerical value indicates an increase in the pain level. In the VAS evaluation, 0 = no pain, 1-4 = mild pain, 5-6 = moderate pain, and 7-10 = severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Nedime Gül DOĞAN ÖZDEMİR, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apaydin Cirik V, Turkmen AS, Ayaz M. Effectiveness of stress ball and relaxation exercises on polymerase chain reaction (RRT-PCR) test-induced fear and pain in adolescents in Turkiye. J Pediatr Nurs. 2023 Jul-Aug;71:135-140. doi: 10.1016/j.pedn.2022.12.001. Epub 2022 Dec 14. PMID 36526480
- [Background] Kocabas P, Khorshid L. A comparison of the effects of a special gynaecological garment and music in reducing the anxiety related to gynaecological examination. J Clin Nurs. 2012 Mar;21(5-6):791-9. doi: 10.1111/j.1365-2702.2011.03958.x. Epub 2011 Dec 15. PMID 22171649
- [Background] Grundstrom H, Wallin K, Bertero C. 'You expose yourself in so many ways': young women's experiences of pelvic examination. J Psychosom Obstet Gynaecol. 2011 Jun;32(2):59-64. doi: 10.3109/0167482X.2011.560692. Epub 2011 Mar 8. PMID 21381979
- [Background] Hilden M, Sidenius K, Langhoff-Roos J, Wijma B, Schei B. Women's experiences of the gynecologic examination: factors associated with discomfort. Acta Obstet Gynecol Scand. 2003 Nov;82(11):1030-6. doi: 10.1034/j.1600-0412.2003.00253.x. PMID 14616277
- [Background] Lin CJ, Chang YC, Chang YH, Hsiao YH, Lin HH, Liu SJ, Chao CA, Wang H, Yeh TL. Music Interventions for Anxiety in Pregnant Women: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2019 Nov 6;8(11):1884. doi: 10.3390/jcm8111884. PMID 31698704
- [Background] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283
- [Background] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915
- [Background] Hudson BF, Ogden J, Whiteley MS. Randomized controlled trial to compare the effect of simple distraction interventions on pain and anxiety experienced during conscious surgery. Eur J Pain. 2015 Nov;19(10):1447-55. doi: 10.1002/ejp.675. Epub 2015 Jan 30. PMID 25641687
- [Background] Yanikkerem E, Ozdemir M, Bingol H, Tatar A, Karadeniz G. Women's attitudes and expectations regarding gynaecological examination. Midwifery. 2009 Oct;25(5):500-8. doi: 10.1016/j.midw.2007.08.006. Epub 2007 Dec 20. PMID 18086509
- [Background] Tugut N, Demirel G, Baser M, Ata EE, Karakus S. Effects of lavender scent on patients' anxiety and pain levels during gynecological examination. Complement Ther Clin Pract. 2017 Aug;28:65-69. doi: 10.1016/j.ctcp.2017.05.006. Epub 2017 May 13. No abstract available. PMID 28779939
- [Background] Haynes AC, Lywood A, Crowe EM, Fielding JL, Rossiter JM, Kent C. A calming hug: Design and validation of a tactile aid to ease anxiety. PLoS One. 2022 Mar 9;17(3):e0259838. doi: 10.1371/journal.pone.0259838. eCollection 2022. PMID 35263344
- [Background] Kurt G, Ozcan NK. The Effect of Virtual Reality On Pain and Anxiety Management During Pelvic Examination: A Randomized Controlled Trial. J Midwifery Womens Health. 2024 Jul-Aug;69(4):543-549. doi: 10.1111/jmwh.13587. Epub 2024 Jan 4. PMID 38178322
- [Background] Henrique AJ, Gabrielloni MC, Rodney P, Barbieri M. Non-pharmacological interventions during childbirth for pain relief, anxiety, and neuroendocrine stress parameters: A randomized controlled trial. Int J Nurs Pract. 2018 Jun;24(3):e12642. doi: 10.1111/ijn.12642. Epub 2018 Mar 7. PMID 29512230
- [Background] Zielinski J, Morawska-Kochman M, Zatonski T. Pain assessment and management in children in the postoperative period: A review of the most commonly used postoperative pain assessment tools, new diagnostic methods and the latest guidelines for postoperative pain therapy in children. Adv Clin Exp Med. 2020 Mar;29(3):365-374. doi: 10.17219/acem/112600. PMID 32129952
- [Background] Manworren RC, Stinson J. Pediatric Pain Measurement, Assessment, and Evaluation. Semin Pediatr Neurol. 2016 Aug;23(3):189-200. doi: 10.1016/j.spen.2016.10.001. Epub 2016 Oct 17. PMID 27989326
- [Background] Spielberger, C. D., Gonzalez-Reigosa, F., Martinez-Urrutia, A., Natalicio, L. F., & Natalicio, D. S. (1971). The state-trait anxiety inventory. Revista Interamericana de Psicologia/Interamerican journal of psychology, 5(3 & 4).
- [Background] Öner, N., & Le Compte, A. (1998). Süreksiz durumluk/sürekli kaygı envanteri el kitabı (2. Baskı). İstanbul: Boğaziçi Üniversitesi, 15-79.